CLINICAL TRIAL: NCT02992262
Title: Ocular Point of Care Ultrasound (POCUS) to Detect Optic Disc Swelling in Comparison to Ophthalmologic Examination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, Director, Research and development unit, Tel-Aviv Medical Center, Israel, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0487-16-TLV
Record Dates: First submitted 2016-12-05; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Papilledema Associated With Increased Intracranial Pressure
MeSH Terms: conditions — Papilledema

INTERVENTIONS:
Device: Point of care ocular ultrasound

SUMMARY:
Pediatric emergency department (PED) physicians frequently encounter children with symptoms that warrant evaluation of the optic disc for suspected increased intracranial pressure (ICP) such as headache, blurred vision, recurrent vomiting etc. Fundoscopic examination, by the PED physician, is considered an essential modality for assessment of the optic disc and the diagnosis of papilledema. Obtaining good visualization of the optic disc requires patient compliance, the ability to open the eyelids, the absence of opacities in the ocular media and a sufficiently large pupillary aperture. Hence, different levels of PED physician training, lack of cooperation, significant ocular or periorbital trauma, contraindications to mydriasis and severe photophobia may hinder direct fundoscopic evaluation.

In the investigators' PED, children requiring fundoscopy are sent to a formal ophthalmologic examination. The investigators aim to evaluate the yield of optic disc height as measured with ocular point of care ultrasound to detect optic disc swelling in comparison to ophthalmologic examination as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients from the PED,
* Aged 0-18 years,
* Who require funduscopic examination and referred to ophthalmologic evaluation.

Exclusion Criteria:

* Direct trauma to the eye with suspicion of ruptured globe or laceration of the eyelid,
* History of glaucoma.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The yield of ocular POCUS in diagnosing optic disc swelling in comparison to ophthalmology evaluation as the gold standard. | Up to 24h from inclusion or until hospital discharge if admitted